CLINICAL TRIAL: NCT03413943
Title: Utilizing Gaze Training to Enhance Laparoscopic Technical Skills Training
Brief Title: Utilizing Gaze Training to Enhance Laparoscopic Skills Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00078782_1
Record Dates: First submitted 2018-01-10; First posted 2018-01-29 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: After identification of the expert gaze, subjects will be randomized into explicit or implicit gaze training techniques.
Who Masked: Participant
Masking Description: The gaze training subjects will be blinded to their cohort assignment, but investigators will know in order to carry out the proper training pending randomization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- explicit gaze training (Experimental): This is an arm of the second phase of the study utilizing gaze training in two different teaching techniques (explicit vs implicit).
  Interventions: Other: gaze training
- implicit gaze training (Experimental): This is an arm of the second phase of the study utilizing gaze training in two different teaching techniques (explicit vs implicit).
  Interventions: Other: gaze training
- sham gaze training (Sham Comparator): This is an arm of the second phase of the study utilizing gaze training in two different teaching techniques (explicit vs implicit).
  Interventions: Other: gaze training

INTERVENTIONS:
Other: gaze training — Gaze training will consist of gaze tracking and then review of performance or the use of an implicit map to train an expert gaze pattern.
  Other Names: Argus Science

SUMMARY:
The purpose of this study is to test the influences of gaze training (GT) on the acquisition of laparoscopic surgical skills. For this purpose, the investigator will compare variants of GT in the second of 2 experiments. These questions will be evaluated using the validated Fundamentals of Laparoscopic Surgery (FLS) module 1, with the overall goal of developing a surgical training curriculum that achieves expert level skill in an expedited timeframe. This research provides a novel approach to general surgery training that has the potential to reduce the amount of time and repetitions required to achieve expert laparoscopic skills.

DETAILED DESCRIPTION:
Developing expert performance requires assessment of the thought processes underlying performance and continued refinement of skills in order to obtain automaticity and intuition. Therefore, developing expert surgical skill is a process likely to take longer than the length of residency, thereby diminishing the quality of care delivered to patients.

The proposed study will implement novel neuroscience technique of gaze training to determine if it has the capacity to accelerate technical surgical skill learning in order to achieve competency and expertise in an earlier timeframe. Studies of skill performance have demonstrated that eye movement patterns can be optimized to improve subsequent motor movements. Therefore, gaze training encourages novices to adopt the more efficient gaze patterns of experts while performing a specific task such as laparoscopic surgery. This technique has been applied in the training of surgical residents in a limited capacity making this project an innovative approach to enhance skill development.

Experiment 2: Determine if gaze training can accelerate the learning of laparoscopic skills.

In this experiment the investigators will first establish expert gaze patterns in the Fundamentals of Laparoscopic Surgery modules 1 and 5 by testing a total of 9 participants, including attending surgeons, senior residents, and novices trained to proficiency. The investigators will then compare behavioral learning curves from non-expert participants without gaze training against those trained using both explicit (by reviewing the expert gaze pattern) and implicit gaze (by using a visual mask during the training, leading the participant to follow the expert gaze) derived from the expert gaze patterns. This will be tested in 3 groups of 20 participants, who train for 40-minutes in each of 6 sessions that occur within 3 weeks.

The investigators hypothesize that both explicit and implicit gaze training will lead to faster skill acquisition, with implicit greater than explicit and measured by trials required to gain proficient module completion scores, relative to the group of participants who practice without any gaze training.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Healthy male and female
* Willing and able to provide informed consent
* Able to follow study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Time to completion | Collected for pre- and post-tests performed prior to and after the 6 separate training sessions within 7-days.
  Completion time for each repetition of FLS task 1

SECONDARY OUTCOMES:
Number of tasks completed | This will be collected for every repetition performed during the 6 separate training sessions within a 7-day period.
  The number of times each FLS task 1 is completed during each training session.
Number of errors | This will be collected for every repetition performed during the 6 separate training sessions within a 7-day period.
  The number of errors (as defined by FLS) during completion of tasks will be recorded and transitioned into a time addition.

CONTACTS AND LOCATIONS:
Overall Officials: Morgan L Cox, MD, Principal Investigator — Duke University; Greg Appelbaum, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Results — https://www.biorxiv.org/content/10.1101/2020.07.17.206763v1